CLINICAL TRIAL: NCT01620645
Title: The Mechanisms of Inflammation and Immunity in COPD and Their Relationship to Exacerbations and Disease Progression.
Brief Title: The MRC/ABPI COPD Cohort v1.7
Acronym: COPDMAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: Royal Free Hampstead NHS Trust (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); Imperial College London (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); University of Sheffield (Other); University Hospitals, Leicester (Other); University of Leicester (Other); University Hospital Birmingham NHS Foundation Trust (Other); University of Birmingham (Other); Cambridge University Hospitals NHS Foundation Trust (Other); University of Cambridge (Other); Liverpool University Hospitals NHS Foundation Trust (Other Government); University of Liverpool (Other); NHS Lothian (Other Government); University of Edinburgh (Other); Newcastle University (Other); University of Nottingham (Other); University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: CSP-83727
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, sputum and urine samples will be collected. Commercially available ELISA assays will be be used to qualify inflammatory markers.
  Quantitative bacterial culture will be performed on sputum samples. Bacterial and viral load will be determined by polymerase chain reaction (PCR). Proteomics such as Cholesterol, BNP, CRP by routine hospital assay techniques. Specific DNA sections will be selected from the genome to identify/confirm genes believed to be associated with different COPD phenotypes by molecular techniques.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- COPD, GOLD II severity or above
  Interventions: Radiation: CT scan and PA chest X-ray

INTERVENTIONS:
Radiation: CT scan and PA chest X-ray — All participants will receive a single high resolution CT scan of the chest. This will be performed using a low tube current, helical technique. Participants may also receive a plain chest X-ray if clinically indicated.
  The total research protocol dose is 2 mSv. The dose from the chest X-ray is insignificant compared with the dose from the CT scan of the chest, therefore all this dose can be considered to be additional to standard of care. A dose of 2 mSv represents a risk of radiation induced detriment of approximately 1 in 10,000 and is equivalent to about 11 months of average natural background radiation in the UK.

SUMMARY:
The UK Medical Research Council (MRC) together with the Association of British Pharmaceutical Industries (ABPI) have recently funded a program designed to foster collaboration between academic COPD researchers and the pharmaceutical industry in the UK, with the aim of developing and furthering our research capacity and expertise for the benefit of patients living with this prevalent and disabling condition. This builds on the strong international track record of COPD research in the UK. The program is divided into four work packages (WP1-4), each with specific aims. WP1 will collate and establish data from patient cohorts and share this information through the development of knowledge management platforms. WP2 will specifically assess how airway micro-organisms impact on COPD and how the effects of bacteria and viruses may be modified. WP3 is concerned with tissue injury and repair which are fundamental processes in the development of COPD. WP4 will examine in detail the potential for improving patient outcomes by targeting the skeletal muscle dysfunction that can profoundly affect exercise capacity.

DETAILED DESCRIPTION:
This study is a multi-centre UK based observational study of a cohort of patients with chronic obstructive pulmonary disease (COPD) funded by the MRC, as part of the MRC/ABPI Inflammation and Immunology Initiative in COPD. This consortium brings together key researchers in the COPD research community with long-standing expertise in understanding bacterial infection, inflammation and immunity.

Understanding the role of bacterial and viral infections, which are often the trigger for exacerbations, and the mechanism of tissue re-modelling and repair following exacerbations is extremely important. Exacerbations and the progression of the disease impose a considerable disability on patients and a financial burden on the health service. In additional, pulmonary inflammation in COPD may result in systemic inflammation. This is associated skeletal muscle dysfunction, as well as worsening other common diseases, such as cardiovascular disease.

We now have a much better understanding of the cellular and molecular mechanisms that underlie COPD and cause the chronic inflammatory process, both locally within the lung and systemically. However, current therapy for COPD is inadequate and relies on long-acting bronchodilators, which do not ameliorate the underlying chronic inflammatory process. Currently available anti-inflammatory therapies are incompletely effective. An improved understanding of the complex mechanisms in COPD is required in order to develop future effective treatments, for which there is a pressing need.

Patients will be recruited from existing cohorts of COPD patients, and indirectly through their general practitioner and outpatient clinics. Patients must have COPD, and all patients will be assessed to ensure the correct diagnosis.

Study patients will be phenotyped by lung morphology and function, biomarkers in blood, sputum and urine, bacterial and viral load in sputum, cardiovascular behaviour, co-morbidities and skeletal muscle function. The patients will be followed up over initially 18 months, with a planned extension to 5 years, to accurately determine the relationship between bacterial and viral infections, tissue re-modelling and skeletal muscle dysfunction with exacerbation frequency and disease progression.

Patients will be phenotyped by:

1. Chest CT-Scan for quantitative measures of lung morphology at baseline
2. ECG and blood pressure to assess cardiovascular risk conferred by systemic inflammation

4)Biomarkers of infection, inflammation and cardiovascular disease in blood, sputum (both spontaneously produced and induced) and urine 5)Quality of life, respiratory symptoms, fatigue, depression, history of cigarette smoking, housing, contact with children and pets and daily activity will be assessed by questionnaire 6)A 6 minute walk test and 4 meter gait speed to determine exercise tolerance and disability 7)Lung function using a spirometer and whole body plethymograph 8)Arterialised blood gases using ear-lobe blood gas analysis 9)Bioimpedance for assessing blood flow and body composition 10)Isometric Muscle strength using quadriceps strain gauge

Patients will be asked to complete a daily diary card on which they will record an increase in two respiratory symptoms, from which we will identify exacerbations, based on our validated criteria of two consecutive days with increase in two symptoms that must include either dyspnoea, sputum purulence or sputum volume. Patients unable to complete the diary cards will be judged incapable of taking part in the research. All patients will provide informed, written consent. Patients will be seen at enrollment, every 6 months thereafter for baseline measurements, at exacerbation and at week 2 and 6 post exacerbation to monitor their recovery.

All patients will undergo a baseline CT scan, at full suspended inspiration with the smallest field of view that includes both lungs. The maximum dose of radiation that each patient with receive from the CT scan is estimated at 2 milli-Sieverts. This is equivalent to about 100 front chest X rays. This compares to an average exposure of 2 milli-Sieverts per year from naturally occurring radioactive material (background radiation). Patients may benefit from detection of previously unknown lung carcinoma and lung abnormalities. At exacerbation visits, some patients may require a chest X-ray as part of standard clinical emergency care e.g. to exclude a pneumothorax or detect pneumonia. The estimated dose of radiation per plain chest X-ray is 0.02 milli-Sieverts.

Blood tests will only be taken by trained personnel. The blood will be analysed for routine haematological parameters, and other body chemicals that might be linked to COPD, ischaemic heart disease and other co-morbridities. The volume of blood taken should not cause any anaemia and routine blood counts will be made to monitor haemoglobin levels.

Both spontaneous and induced sputum specimens will be taken. The induced sputum may cause coughing and some shortness of breath. Patients will be closely monitored and their lung function checked to ensure their safety. We have previously shown that induced sputum sampling is a safe procedure in COPD.

Patients will be asked to walk for 6 minutes and the distance recorded. Patients heart rate and oxygen saturation will be monitored before and after the walk. Patients may experience shortness of breath during this test. Supplementary oxygen will be available if the patient desaturates during the test. Additional assessment of muscle strength and disability will be carried out using a quadriceps strain gauge, the four meter gait speed test and the short physical performance battery. The patient should not experience any more dyspnoea than they would normally encounter in everyday life and the quadriceps strain gauge will only be performed if there are no underlying musculoskeletal or neurological contra-indications.

Some investigations described above are specific to certain centres collaborating in this study and not all tests will be performed on all patients. The tests which will be requested for each individual patient will be fully explained during their initial visit at the appropriate study site.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed spirometric evidence of moderate to very severe COPD (stage II to IV) according to the WHO GOLD criteria:
* All patients FEV1/FVC <70%
* Stage II FEV1 50-80% predicted
* Stage III FEV1 30-50% predicted
* Stage IV FEV1 <30% predicetd or <50% predicted and chronic respiratory symptoms
* Past or present smokers
* Gender: male or female
* Age >40 years at recruitment
* Reasonable command of English to complete daily diary cards

Exclusion Criteria:

* History of asthma
* History of neoplasia
* History of other significant respiratory disease
* Pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from existing cohorts and may have participated in previously approved studies.
  Potential primary care patients will be identified from databases held in practices and contacted, by the GP, by letter in the first instance. If the patient replies to the GP that they are willing to participate in the research, then a telephone call will be made by the research team to arrange a clinic visit.
  Potential outpatient participants will be identified by the outpatient respiratory physician and if willing to participate will be referred to the research team via telephone call or referral letter.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-02

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Free Hampstead NHS Trust, London, London, United Kingdom

REFERENCES:
- [Derived] Wang Z, Singh R, Miller BE, Tal-Singer R, Van Horn S, Tomsho L, Mackay A, Allinson JP, Webb AJ, Brookes AJ, George LM, Barker B, Kolsum U, Donnelly LE, Belchamber K, Barnes PJ, Singh D, Brightling CE, Donaldson GC, Wedzicha JA, Brown JR; COPDMAP. Sputum microbiome temporal variability and dysbiosis in chronic obstructive pulmonary disease exacerbations: an analysis of the COPDMAP study. Thorax. 2018 Apr;73(4):331-338. doi: 10.1136/thoraxjnl-2017-210741. Epub 2017 Dec 21. PMID 29269441